CLINICAL TRIAL: NCT05387291
Title: Effectiveness of the Application of a Nursing Intervention Program in the Management of Parental Anxiety and Infant Pain in the Surgical Process of Children to be Circumcised
Brief Title: Nursing Intervention Program in the Management of Parental Anxiety and Infant Pain in the Surgical Process of Children to be Circumcised
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Girona (Other)
Responsible Party: Principal Investigator, Lyudmila Andrusenko Kalchenko, Principal Investigator, Universitat de Girona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2022-05-12; First posted 2022-05-24 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Anxiety; Pain, Postoperative; Child Development
Keywords: Anxiety; Child Preschool; Circumcision Male; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative; Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to one group (intervention) or the other (control).
Who Masked: Participant
Masking Description: The subjects do not know which group they are in, as some are given the usual intervention (control group) and others the intervention (intervention group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nursing Intervention (Experimental): The intervention group will undergo an education program related to the circumcision process for the child's relatives/guardians.
  Interventions: Behavioral: Intervention group
- Usual intervention (Other): The control group will receive the usual intervention of the center.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Intervention group — The intervention group will undergo an education program related to the circumcision process for the child's relatives/guardians.
  Arms: Nursing Intervention
Behavioral: Control group — The control group will receive the usual intervention of the center.
  Arms: Usual intervention

SUMMARY:
Entering the hospital and waiting for surgery is a very stressful time for people. According to some studies, surgical interventions in children generate in family members concerns related to: anesthesia, fear of being harmed, penile injury, excessive pain, the death of their child, not being able to contain their own anxiety and, therefore, participants may have difficulties in assuming an active role in caring for their child .

For these reasons, the investigators propose the development and implementation of an action program for the reduction of child pain and anxiety in parents in the foreign Muslim population residing in Spain.

DETAILED DESCRIPTION:
1. Introduction Entering the hospital and waiting for surgery is a very stressful time for people. According to some studies, surgical interventions in children generate in family members concerns related to: anesthesia, fear of being harmed, penile injury, excessive pain, the death of their child, not being able to contain their own anxiety and, therefore, participants may have difficulties in assuming an active role in caring for their child.

   For these reasons, the investigators propose the development and implementation of an action program for the reduction of child pain and anxiety in parents in the foreign Muslim population residing in Spain.
2. Hypothesis / problem A nursing intervention program in the surgical process of circumcision decreases the degree of anxiety of family members and reduces infant pain.
3. Methodology A randomized clinical trial will be carried out at the Policlínica Maresme, located in Pineda de Mar, on the relatives/guardians and children aged 0-3 years who are going to undergo circumcision.

The intervention group will undergo an education program related to the circumcision process for the child's relatives/guardians. The control group will receive the usual intervention of the center. It has been estimated that 157 subjects are needed in each group, estimating a loss to follow-up of 10%.

Among other variables, the preoperative anxiety level of the parents will be measured using the Hamilton scale; intraoperatively, child pain will be measured using the FLACC scale and, subsequently, a postoperative telephone follow-up will be carried out during the 2 and 10 days following the intervention, to assess aspects related to the clinical evolution of the surrounded child and the resolution of any doubts that the caregivers may have.

The confidentiality of the study participants will be guaranteed. The research project has been approved by the Comité d'Ètica d'Investigació Clínica amb Medicaments de l'Hospital de Mataró with code CEIm 03/22.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-3 years who are going to undergo circumcision and the relatives/guardians.

Exclusion Criteria:

* Children with micropenis

Ages: 0 Months to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-12 (Actual); Study Completion 2022-05-22 (Actual)

PRIMARY OUTCOMES:
Preoperative anxiety level of the parents | Preoperative phase
  The preoperative anxiety level of the parents will be measured using the Hamilton scale. Minimum value 0, Maximum value 56. The higher the score, the higher the anxiety.
Intraoperatively Pain Child | Intraoperatively Phase
  Child pain will be measured using the Face, Legs, Activity, Cry, Consolability scale (FLACC scale). Minimum value 0, Maximum value 10. The higher the score, the higher the pain.

SECONDARY OUTCOMES:
Postoperative telephone follow-up | Days 2 and 10 after the intervention.
  Postoperative telephone follow-up will be carried out to assess aspects related to the clinical evolution of the surrounded child and the resolution of any doubts that the caregivers may have.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlínica Maresme, Pineda de Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
The data will only be used by the study investigators.